CLINICAL TRIAL: NCT00908830
Title: Pharmacokinetics of Mycophenolic Acid in Cystic Fibrosis Lung Transplant Recipients
Brief Title: Effects of Mycophenolate Mofetil in Cystic Fibrosis Lung Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tammy Ojo Clark, MD, Assistant Professor of Internal Medicine, University of Michigan
Other Study IDs: UM 20989
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis; Lung Transplant
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cystic fibrosis: Lung transplant patients with cystic fibrosis. Measuring MPA levels in cystic fibrosis lung transplant patients for pharmacokinetic parameters.
- Non-cystic fibrosis lung transplant: Non-cystic fibrosis lung transplant patients. Non-cystic fibrosis lung transplant patients will have MPA levels drawn after their dose to determine pharmacokinetic parameters.

SUMMARY:
Lung transplantation is a life saving procedure for patients with a terminal lung disease such as cystic fibrosis. Approximately, one in 3,500 children in the United States are born with cystic fibrosis each year with the predicted survival reaching 36.9 years in 2006. Cystic fibrosis was the third lead indication for lung transplantation in 2006. Cystic fibrosis is a genetic disease that can affect the way the body can remove salt from various organs. It results in mucus blocking the ducts of the lungs and pancreas leading to inability to handle oxygen and malabsorption of nutrients. Malabsorption is a common complication of cystic fibrosis that can affect the way the anti-rejection medications are absorbed. One medication that is utilized after transplant to prevent rejection is mycophenolate mofetil. This medication may not be absorbed adequately in this population due to their disease thus placing these patients at increased risk of rejection. At the investigators' institution, all transplant patients are initiated at the same mycophenolate dose regardless of their underlying disease. The limited available literature regarding cystic fibrosis transplant patients and mycophenolate suggests that these patients require higher doses due to their erratic absorption. The purpose of this study is to evaluate the effects of mycophenolate mofetil on the body in lung transplant patients who have cystic fibrosis in efforts to improve survival outcomes.

DETAILED DESCRIPTION:
Background:

Lung transplantation has been established as a viable treatment for cystic fibrosis (CF) patients who have end-stage lung disease. CF is a genetic disorder which is caused by mutations in the cystic fibrosis transmembrane conductance regulator gene. These mutations cause abnormal transport of sodium chloride which affects various organs. In the lungs, there is a reduction in mucociliary clearance leading to viscous mucus that can block the airways. In addition to obstruction of the airways, the stagnant mucus provides a good medium for microorganisms leading to infectious complications.1,2 Approximately one in 3,500 children in the United States are born with CF each year with the predicted survival reaching 36.9 years in 2006.3 CF was the third leading indication (16%) for lung transplantation in 2006.4

The success of transplantation has been due to the advances in immunosuppression over the years. Within the past ten years, the substantial changes in the immunosuppression regimen include more transplant centers utilizing induction therapy (29% vs. 50% in 1995 and 2004, respectively); and baseline immunosuppression shifted from cyclosporine-based in 1995 (77%) to tacrolimus-based in 2004 (70%).5 In addition, mycophenolate mofetil (MMF) has been replacing azathioprine as the purine synthesis antagonist in maintenance regimens in the recent years.4

Gastrointestinal malabsorption is a common complication of CF that can affect the impact of immunosuppression. It has been shown that CF patients can have sub-therapeutic calcineurin inhibitors.6,7 However, little information regarding MMF pharmacokinetics (PK) exist in this population. One small observational study of 30 stable lung-transplant recipients demonstrated that the CF patients (n=7) required at least 30% higher doses to achieve similar pre-dose levels of mycophenolic acid (MPA) to that of non-CF patients (n=6).8 The authors did not include any other PK parameters in their results. In a second study, 12-hour PK of MPA and its glucuronide metabolites were characterized in 21 stable lung transplant recipients. The authors included 5 CF patients and found no significant difference in PK parameters except for the ratio of MPA glucuronide and MPA (MPAG/MPA) between the CF and non-CF patients. However, the CF patients tended to have a lower area under the curve (AUC) than non-CF patients. Inter- or intra-patient variability of MPA AUC was not determined in this study.9 In addition, these previous studies did not distinguish tacrolimus-based regimen from cyclosporine-based regimen.

At our institution, CF patients are managed the same as any other lung transplant patients in regards to immunosuppression. Standard starting dose for MMF is 1000mg twice daily within our institution, and pre-dose MPA levels are not routinely measured since they do not reflect MPA exposure. In contrast, other transplant centers dose MMF higher in CF patients based on the limited reports above. The purpose of this study is to determine PK of MPA and MPAG in CF patients on tacrolimus and compare them to a cohort of non-CF lung transplant patients.

Outline of the study:

We will conduct an open-label, PK study in stable CF lung transplant patients. Our study will also evaluate non-CF patients as the control group. Each patient will have three biweekly PK study visits. On the PK study days, patients will be admitted to the Michigan Clinical Research Unit (MCRU) at the University of Michigan Health Center. After administration of morning dose of MMF, serial blood samples will be collected at the following time intervals: immediately before and 0.5, 1, 1.5, 2, 4, 6, 9, and 12 hours after dosing. Serum creatinine and serum albumin will also be drawn. Vial of blood will be also collected to measure the function of IMPDH. Standardized meals will be provided on PK study days. Serum concentrations of total MPA and MPAG will be determined by a validated liquid chromatography with tandem mass spectrometry method.10

Outcome Measures:

Pharmacokinetic parameters of MPA and MPAG will be determined by noncompartmental methods. The area under the plasma concentration-time curve from time 0 to 12 hours (AUC) will be calculated by the trapezoidal rule. Maximum serum concentration (Cmax) and time to reach Cmax (Tmax) will be determined from visual inspection of the concentration-time profile. Clearance (CL/F) will be calculated by dose divided by AUC. Samples will be obtained to measure IMPDH and correlated with PK parameters. These tests will be assayed by Les Shaw at the University of Pennsylvania.

Statistical Analysis and Sample Size All PK parameters will be reported as mean and standard deviation. To analyze the inter- and intra-patient variability, coefficients of variation of the MPA AUC's will be calculated. Differences in the variables between the CF and non-CF patients will be determined by Student's t-test or Wilcoxon signed rank test. A two-sided p-value less than 0.05 will be considered significant.

Our sample size will be five CF and non-CF lung transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide informed consent and be compliant with the study procedures
* Between 18-70 years of age
* Greater than 1 year post-transplant
* Have no evidence of acute rejection at 1 year post-transplant biopsy or within three months of study entry
* Stable mycophenolate mofetil dose
* Stable renal function

Exclusion Criteria:

* Serum creatinine greater than 2 mg/dl
* Received pulse steroids within 3 months of the study entry
* Chronic diarrhea
* Concurrently on interacting medications (cholestyramine, etc)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients with and without cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Ojo, MD, Principal Investigator — University of Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystic Fibrosis: Lung transplant patients with cystic fibrosis. Measuring MPA levels in cystic fibrosis lung transplant patients for pharmacokinetic parameters.
  mycophenolate mofetil : Patients will take their own 500-mg tablets of mycophenolate mofetil
- Non-cystic Fibrosis Lung Transplant: Non-cystic fibrosis lung transplant patients. Non-cystic fibrosis lung transplant patients will have MPA levels drawn after their dose to determine pharmacokinetic parameters.
  mycophenolate mofetil : Patients will take their own 500-mg tablets of mycophenolate mofetil
Period: Overall Study
Arm/Group | Cystic Fibrosis | Non-cystic Fibrosis Lung Transplant
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis | Non-cystic Fibrosis Lung Transplant | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (6.8) | 59.4 (9.0) | 45.0 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Pharmacokinetics of Mycophenolic Acid and Mycophenolic Acid Glucuronide in Stable Cystic Fibrosis and Non-Cystic Fibrosis Lung Transplant Recipients.
Description: The AUC is the area under the concentration-time curve from time 0 to 12 hours. The AUC is measured in units of micrograms of mycophenolic acid (MPA) per milliliter of plasma (mcg/mL) multiplied by time in hours (mg*h/L) and in units of micrograms of mycophenolic acid glucuronide (MPAG) per milliliter of plasma (mcg/mL) multiplied by time in hours (mg*h/L). Apparent oral clearance (CL/F) was calculated by dose/AUC0-12.
Time Frame: 0 hours pre-dose and again at 0.5, 1, 1.5, 2, 4, 6, 9, and 12 hours post-dose
Measure: Mean (Standard Error); unit: mg*h/L
Arm/Group | Cystic Fibrosis | Non-cystic Fibrosis Lung Transplant
Number analyzed (Participants) | 5 | 5
mg*h/L
  MPA AUC | 47.7 (13.7) | 83.1 (27.9)
  MPAG AUC | 569 (204) | 911 (249)

2. Secondary Outcome: Inter- and Intra-patient Variability of Mycophenolic Acid Exposure (AUC) in Cystic Fibrosis Lung Transplant Recipients on Tacrolimus Based Immunosuppression.
Description: Inter- and intra-patient variability will be calculated by the coefficients of variation (CV) of the MPA AUC (mg*h/L).
  To analyze the intra- and interindividual variability, the coefficient of variation (CV) was calculated by dividing the standard deviation by the mean of the PK parameters from the 3 PK visits and the 5 study patients in each group, respectively. Inter-individual CVs presented are only comparing within the individuals per arm, not across or between arms.
Time Frame: 0 hours pre-dose and again at 0.5, 1, 1.5, 2, 4, 6, 9, and 12 hours post-dose
Measure: Mean (Standard Deviation); unit: percent CV
Arm/Group | Cystic Fibrosis | Non-cystic Fibrosis Lung Transplant
Number analyzed (Participants) | 5 | 5
percent CV
  MPA AUC..Intraindividual | 16.6 (6.1) | 13.8 (5.3)
  MPA AUC..Interindividual | 31.2 (1.5) | 36.3 (5.6)
  MPAG AUC..Intraindividual | 16.6 (6.5) | 15.9 (6.7)
  MPAG AUC..Interindividual | 37.3 (6.1) | 27.8 (3.2)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Cystic Fibrosis | Non-cystic Fibrosis Lung Transplant
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Since a comparative PK study with intravenous MMF was not conducted in our cohorts, the reason for the differences observed in the PK parameters between the 2 cohorts remains unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes